CLINICAL TRIAL: NCT04488575
Title: A Phase 2 Double-blind Placebo-controlled Study Investigating the Safety and Efficacy of EDP1815 in the Treatment of Patients Hospitalized With SARS-CoV-2 Infection
Brief Title: Safety and Efficacy of EDP1815 in the Treatment of Patients Hospitalized With COVID-19 Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient study defined patient population
Sponsor: Evelo Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EDP1815-205
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-07

CONDITIONS: Covid19
Keywords: SARS-CoV-2; corona virus; coronavirus; corona
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either the active (EDP1815) or placebo group (1:1 randomization), in addition to standard of care. Dosing will be initiated on a twice daily regime for the first 3 days (6 doses) and then once daily for the remaining 11 days (14 days total treatment course).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Fully blinded to the participants, investigator, and sponsor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EDP1815 (Experimental): Patients will receive EDP1815 in addition to standard of care
  Interventions: Drug: EDP1815
- Placebo (Placebo Comparator): Patients will receive placebo in addition to standard of care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP1815 — EDP1815 is an orally administered monoclonal microbe
  Arms: EDP1815
Drug: Placebo — Placebo oral capsule
  Arms: Placebo

SUMMARY:
Evelo will investigate the safety and efficacy of EDP1815 in the treatment of patients hospitalized with SARS-CoV-2 Infection

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled clinical study to assess the safety and efficacy of EDP1815 in patients hospitalized with COVID-19 infection.

The study is designed to evaluate the efficacy of EDP1815 at reducing time to resolution of symptoms, preventing progression of COVID-19 symptoms and preventing COVID-Related Complications (CRC)

ELIGIBILITY:
Key Inclusion Criteria:

1. Hospitalized within the last 36 hours.
2. Receiving any form of supplementary oxygen therapy at baseline.
3. Confirmed COVID-19 viral infection by RTPCR at screening.
4. Age:

   1. 18-65 years old, OR
   2. >65 year-olds can be included after Data Monitoring Committee (DMC) approval

Key Exclusion Criteria:

1. Contraindications/hypersensitivity to P histicola or any of the capsule excipients
2. Patients with chronic hypoxia or underlying significant chronic respiratory disease (such as Chronic Obstructive Pulmonary Disease (COPD), Pulmonary Fibrosis, or Bronchiectasis).
3. Admission to ICU at time of screening.
4. Mechanically ventilated, on continuous positive airway pressure (CPAP), or on non-invasive ventilation at the time of screening.
5. Patient is taking a systemic immunosuppressive agent such as, but not limited to, oral steroids, methotrexate, azathioprine, ciclosporin, or tacrolimus, unless these are given as part of COVID standard of care treatment.
6. Patient has a diagnosed primary immunodeficiency.
7. Patient has a diagnosis of HIV/AIDS
8. Patient has pre-existing known chronic kidney disease stage 4 or 5 or requiring renal replacement therapy (i.e. estimated glomerular filtration rate (eGFR) <30ml/min/1.73m2)
9. Patient has pre-existing known significant liver disease with Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 5.0 x upper limit of normal (ULN)
10. Patient has pre-existing known significant gastrointestinal tract disease expected to affect absorption within the small intestine (e.g. short bowel syndrome, inflammatory bowel disease affecting the small intestine, gastroparesis); or prior malabsorptive bariatric surgery that could interfere with GI delivery and transit time.
11. GI signs or symptoms equivalent to CTCAE v5.0, gastrointestinal disorders, grade 3 or 4 event.
12. Patient has pre-existing known substantially impaired cardiac function or pre-existing clinically significant cardiac diseases, including unstable angina or acute myocardial infarction ≤ 6 weeks prior to Screening.
13. Currently participating in an interventional clinical trial (observational studies allowed).
14. Moribund at time of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-05-16 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Reynold Panettieri, MD, Principal Investigator — Rutgers, The State University of New Jersey; Douglas Maslin, MD, Study Director — Evelo Biosciences
Locations (4):
- United States (3):
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - The University Hospital, Newark, New Jersey
  - DHR Health Institute, Edinburg, Texas
- Hacettepe University Adult Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | EDP1815
Started | 7 | 9
Completed | 7 | 4
Not Completed | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | EDP1815 | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 8 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the Lowest S/F Oxygen Ratio in Days 1 to 14
Description: Worst pulmonary function as measured by the change in Oxygen Saturation (SpO2) / Fraction of Inspired Oxygen (FiO2) [S/F ratio]
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Ratio | -30.0 (114.95) | -63.8 (76.85)

2. Secondary Outcome: Change in S/F Ratio
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using change in S/F ratio at days 4, 7, 10 and 14/discharge day.
Time Frame: 14 days
Population: All participants providing data at the relevant timepoints.
Measure: Mean (Full Range); unit: Ratio
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Ratio
  Day 4: number analyzed (Participants) | 7 | 8
  Day 4 | 37.4 [-59.0 to 148.0] | -23.0 [-188.0 to 167.0]
  Day 7: number analyzed (Participants) | 3 | 3
  Day 7 | -16.0 [-65.0 to 20.0] | -86.7 [-130.0 to 6.0]
  Day 10: number analyzed (Participants) | 2 | 2
  Day 10 | 37.0 [-68.0 to 142.0] | -111.0 [-115.0 to -107.0]
  Day 14: number analyzed (Participants) | 1 | 2
  Day 14 | -83.0 [-83.0 to -83.0] | -14.0 [-53.0 to 25.0]

3. Secondary Outcome: Percentage Change in S/F Ratio
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using percentage change in S/F ratio at days 4, 7, 10 and 14/discharge day.
Time Frame: 14 days
Population: All participants providing data at the relevant timepoints.
Measure: Mean (Full Range); unit: percentage change
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
percentage change
  Day 4: number analyzed (Participants) | 7 | 8
  Day 4 | 10.97 [-33.1 to 49.3] | -5.33 [-66.0 to 104.4]
  Day 7: number analyzed (Participants) | 3 | 3
  Day 7 | -10.41 [-36.5 to 8.4] | -36.48 [-57.6 to 2.1]
  Day 10: number analyzed (Participants) | 2 | 2
  Day 10 | 109.7 [-38.2 to 147.9] | -46.6 [-48.7 to -44.4]
  Day 14: number analyzed (Participants) | 1 | 2
  Day 14 | -46.6 [-46.6 to -46.6] | -5.7 [-22.0 to 10.6]

4. Secondary Outcome: Percentage of Participants at Each Level on the WHO OSCI Score
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using percentage of participants at each level on the WHO OSCI score at days 4, 7, 14, 21 and 42.
  (WHO OSCI - World health Organization, Ordinal Scale for Clinical Improvement; 0=unifected - 8=death)
Time Frame: 42 days
Population: All participants providing data at the relevant timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Participants
  Day 4: WHO OSCI score - 0 | 1 | 0
  Day 4: WHO OSCI score - 1 | 0 | 0
  Day 4: WHO OSCI score - 2 | 0 | 1
  Day 4: WHO OSCI score - 3 | 1 | 1
  Day 4: WHO OSCI score - 4 | 5 | 5
  Day 4: WHO OSCI score - 5 | 0 | 1
  Day 4: WHO OSCI score - 6 | 0 | 1
  Day 4: WHO OSCI score - 7 | 0 | 0
  Day 4: WHO OSCI score - 8 | 0 | 0
  Day 7: number analyzed (Participants) | 7 | 5
  Day 7: WHO OSCI score - 0 | 1 | 0
  Day 7: WHO OSCI score - 1 | 0 | 0
  Day 7: WHO OSCI score - 2 | 3 | 2
  Day 7: WHO OSCI score - 3 | 0 | 0
  Day 7: WHO OSCI score - 4 | 2 | 1
  Day 7: WHO OSCI score - 5 | 1 | 1
  Day 7: WHO OSCI score - 6 | 0 | 1
  Day 7: WHO OSCI score - 7 | 0 | 0
  Day 7: WHO OSCI score - 8 | 0 | 0
  Day 14: number analyzed (Participants) | 6 | 6
  Day 14: WHO OSCI score - 0 | 3 | 1
  Day 14: WHO OSCI score - 1 | 0 | 0
  Day 14: WHO OSCI score - 2 | 2 | 3
  Day 14: WHO OSCI score - 3 | 0 | 0
  Day 14: WHO OSCI score - 4 | 1 | 1
  Day 14: WHO OSCI score - 5 | 0 | 0
  Day 14: WHO OSCI score - 6 | 0 | 1
  Day 14: WHO OSCI score - 7 | 0 | 0
  Day 14: WHO OSCI score - 8 | 0 | 0
  Day 21: number analyzed (Participants) | 6 | 6
  Day 21: WHO OSCI score - 0 | 4 | 1
  Day 21: WHO OSCI score - 1 | 0 | 0
  Day 21: WHO OSCI score - 2 | 1 | 4
  Day 21: WHO OSCI score - 3 | 0 | 0
  Day 21: WHO OSCI score - 4 | 1 | 0
  Day 21: WHO OSCI score - 5 | 0 | 0
  Day 21: WHO OSCI score - 6 | 0 | 1
  Day 21: WHO OSCI score - 7 | 0 | 0
  Day 21: WHO OSCI score - 8 | 0 | 0
  Day 42: number analyzed (Participants) | 5 | 3
  Day 42: WHO OSCI score - 0 | 4 | 3
  Day 42: WHO OSCI score - 1 | 0 | 0
  Day 42: WHO OSCI score - 2 | 0 | 0
  Day 42: WHO OSCI score - 3 | 0 | 0
  Day 42: WHO OSCI score - 4 | 1 | 0
  Day 42: WHO OSCI score - 5 | 0 | 0
  Day 42: WHO OSCI score - 6 | 0 | 0
  Day 42: WHO OSCI score - 7 | 0 | 0
  Day 42: WHO OSCI score - 8 | 0 | 0

5. Secondary Outcome: Percentage of Participants With Shifts From Each Level of the WHO OSCI Score at Baseline
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using percentage of participants with shifts from each level of the WHO OSCI score at baseline at days 4, 7, 14, 21 and 42.
  (WHO OSCI - World health Organization, Ordinal Scale for Clinical Improvement; 0=uninfected - 8=death)
Time Frame: 42 days
Population: All participants providing data at the relevant timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Participants
  Day 4: Baseline WHO OSCI score 4; WHO OSCI Score - 0 | 1 | 0
  Day 4: Baseline WHO OSCI score 4; WHO OSCI Score - 1 | 0 | 0
  Day 4: Baseline WHO OSCI score 4; WHO OSCI Score - 2 | 0 | 1
  Day 4: Baseline WHO OSCI score 4; WHO OSCI Score - 3 | 1 | 1
  Day 4: Baseline WHO OSCI score 4; WHO OSCI Score - 4 | 4 | 5
  Day 4: Baseline WHO OSCI score 4; WHO OSCI Score - 5 | 0 | 1
  Day 4: Baseline WHO OSCI score 4; WHO OSCI Score - 6 | 0 | 1
  Day 4: Baseline WHO OSCI score 4; WHO OSCI Score - 7 | 0 | 0
  Day 4: Baseline WHO OSCI score 4; WHO OSCI Score - 8 | 0 | 0
  Day 4: Baseline WHO OSCI score 5; WHO OSCI Score - 0 | 0 | 0
  Day 4: Baseline WHO OSCI score 5; WHO OSCI Score - 1 | 0 | 0
  Day 4: Baseline WHO OSCI score 5; WHO OSCI Score - 2 | 0 | 0
  Day 4: Baseline WHO OSCI score 5; WHO OSCI Score - 3 | 0 | 0
  Day 4: Baseline WHO OSCI score 5; WHO OSCI Score - 4 | 1 | 0
  Day 4: Baseline WHO OSCI score 5; WHO OSCI Score - 5 | 0 | 0
  Day 4: Baseline WHO OSCI score 5; WHO OSCI Score - 6 | 0 | 0
  Day 4: Baseline WHO OSCI score 5; WHO OSCI Score - 7 | 0 | 0
  Day 4: Baseline WHO OSCI score 5; WHO OSCI Score - 8 | 0 | 0
  Day7: number analyzed (Participants) | 7 | 5
  Day7: Baseline WHO OSCI score 4; WHO OSCI Score - 0 | 1 | 0
  Day7: Baseline WHO OSCI score 4; WHO OSCI Score - 1 | 0 | 0
  Day7: Baseline WHO OSCI score 4; WHO OSCI Score - 2 | 3 | 2
  Day7: Baseline WHO OSCI score 4; WHO OSCI Score - 3 | 0 | 0
  Day7: Baseline WHO OSCI score 4; WHO OSCI Score - 4 | 1 | 1
  Day7: Baseline WHO OSCI score 4; WHO OSCI Score - 5 | 1 | 1
  Day7: Baseline WHO OSCI score 4; WHO OSCI Score - 6 | 0 | 1
  Day7: Baseline WHO OSCI score 4; WHO OSCI Score - 7 | 0 | 0
  Day7: Baseline WHO OSCI score 4; WHO OSCI Score - 8 | 0 | 0
  Day7: Baseline WHO OSCI score 5; WHO OSCI Score - 0 | 0 | 0
  Day7: Baseline WHO OSCI score 5; WHO OSCI Score - 1 | 0 | 0
  Day7: Baseline WHO OSCI score 5; WHO OSCI Score - 2 | 0 | 0
  Day7: Baseline WHO OSCI score 5; WHO OSCI Score - 3 | 0 | 0
  Day7: Baseline WHO OSCI score 5; WHO OSCI Score - 4 | 1 | 0
  Day7: Baseline WHO OSCI score 5; WHO OSCI Score - 5 | 0 | 0
  Day7: Baseline WHO OSCI score 5; WHO OSCI Score - 6 | 0 | 0
  Day7: Baseline WHO OSCI score 5; WHO OSCI Score - 7 | 0 | 0
  Day7: Baseline WHO OSCI score 5; WHO OSCI Score - 8 | 0 | 0
  Day 14: number analyzed (Participants) | 6 | 6
  Day 14: Baseline WHO OSCI score 4; WHO OSCI Score - 0 | 3 | 1
  Day 14: Baseline WHO OSCI score 4; WHO OSCI Score - 1 | 0 | 0
  Day 14: Baseline WHO OSCI score 4; WHO OSCI Score - 2 | 2 | 3
  Day 14: Baseline WHO OSCI score 4; WHO OSCI Score - 3 | 0 | 0
  Day 14: Baseline WHO OSCI score 4; WHO OSCI Score - 4 | 1 | 1
  Day 14: Baseline WHO OSCI score 4; WHO OSCI Score - 5 | 0 | 0
  Day 14: Baseline WHO OSCI score 4; WHO OSCI Score - 6 | 0 | 1
  Day 14: Baseline WHO OSCI score 4; WHO OSCI Score - 7 | 0 | 0
  Day 14: Baseline WHO OSCI score 4; WHO OSCI Score - 8 | 0 | 0
  Day 14: Baseline WHO OSCI score 5; WHO OSCI Score - 0 | 0 | 0
  Day 14: Baseline WHO OSCI score 5; WHO OSCI Score - 1 | 0 | 0
  Day 14: Baseline WHO OSCI score 5; WHO OSCI Score - 2 | 0 | 0
  Day 14: Baseline WHO OSCI score 5; WHO OSCI Score - 3 | 0 | 0
  Day 14: Baseline WHO OSCI score 5; WHO OSCI Score - 4 | 0 | 0
  Day 14: Baseline WHO OSCI score 5; WHO OSCI Score - 5 | 0 | 0
  Day 14: Baseline WHO OSCI score 5; WHO OSCI Score - 6 | 0 | 0
  Day 14: Baseline WHO OSCI score 5; WHO OSCI Score - 7 | 0 | 0
  Day 14: Baseline WHO OSCI score 5; WHO OSCI Score - 8 | 0 | 0
  Day 21: number analyzed (Participants) | 6 | 6
  Day 21: Baseline WHO OSCI score 4; WHO OSCI Score - 0 | 4 | 1
  Day 21: Baseline WHO OSCI score 4; WHO OSCI Score - 1 | 0 | 0
  Day 21: Baseline WHO OSCI score 4; WHO OSCI Score - 2 | 1 | 4
  Day 21: Baseline WHO OSCI score 4; WHO OSCI Score - 3 | 0 | 0
  Day 21: Baseline WHO OSCI score 4; WHO OSCI Score - 4 | 1 | 0
  Day 21: Baseline WHO OSCI score 4; WHO OSCI Score - 5 | 0 | 0
  Day 21: Baseline WHO OSCI score 4; WHO OSCI Score - 6 | 0 | 1
  Day 21: Baseline WHO OSCI score 4; WHO OSCI Score - 7 | 0 | 0
  Day 21: Baseline WHO OSCI score 4; WHO OSCI Score - 8 | 0 | 0
  Day 21: Baseline WHO OSCI score 5; WHO OSCI Score - 0 | 0 | 0
  Day 21: Baseline WHO OSCI score 5; WHO OSCI Score - 1 | 0 | 0
  Day 21: Baseline WHO OSCI score 5; WHO OSCI Score - 2 | 0 | 0
  Day 21: Baseline WHO OSCI score 5; WHO OSCI Score - 3 | 0 | 0
  Day 21: Baseline WHO OSCI score 5; WHO OSCI Score - 4 | 0 | 0
  Day 21: Baseline WHO OSCI score 5; WHO OSCI Score - 5 | 0 | 0
  Day 21: Baseline WHO OSCI score 5; WHO OSCI Score - 6 | 0 | 0
  Day 21: Baseline WHO OSCI score 5; WHO OSCI Score - 7 | 0 | 0
  Day 21: Baseline WHO OSCI score 5; WHO OSCI Score - 8 | 0 | 0
  Day 42: number analyzed (Participants) | 5 | 3
  Day 42: Baseline WHO OSCI score 4; WHO OSCI Score - 0 | 4 | 3
  Day 42: Baseline WHO OSCI score 4; WHO OSCI Score - 1 | 0 | 0
  Day 42: Baseline WHO OSCI score 4; WHO OSCI Score - 2 | 0 | 0
  Day 42: Baseline WHO OSCI score 4; WHO OSCI Score - 3 | 0 | 0
  Day 42: Baseline WHO OSCI score 4; WHO OSCI Score - 4 | 1 | 0
  Day 42: Baseline WHO OSCI score 4; WHO OSCI Score - 5 | 0 | 0
  Day 42: Baseline WHO OSCI score 4; WHO OSCI Score - 6 | 0 | 0
  Day 42: Baseline WHO OSCI score 4; WHO OSCI Score - 7 | 0 | 0
  Day 42: Baseline WHO OSCI score 4; WHO OSCI Score - 8 | 0 | 0
  Day 42: Baseline WHO OSCI score 5; WHO OSCI Score - 0 | 0 | 0
  Day 42: Baseline WHO OSCI score 5; WHO OSCI Score - 1 | 0 | 0
  Day 42: Baseline WHO OSCI score 5; WHO OSCI Score - 2 | 0 | 0
  Day 42: Baseline WHO OSCI score 5; WHO OSCI Score - 3 | 0 | 0
  Day 42: Baseline WHO OSCI score 5; WHO OSCI Score - 4 | 0 | 0
  Day 42: Baseline WHO OSCI score 5; WHO OSCI Score - 5 | 0 | 0
  Day 42: Baseline WHO OSCI score 5; WHO OSCI Score - 6 | 0 | 0
  Day 42: Baseline WHO OSCI score 5; WHO OSCI Score - 7 | 0 | 0
  Day 42: Baseline WHO OSCI score 5; WHO OSCI Score - 8 | 0 | 0

6. Secondary Outcome: Number of Participants Remaining at Their Baseline Score on the WHO OSCI (or Lower)
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using percentage of participants remaining at their baseline score on the WHO OSCI (or lower) at days 4, 7, 14, 21 and 42. Once a participant has increased their WHO OSCI score they are not considered to have remained at or below their baseline value at future visits regardless of whether their score returns to or below their baseline value.
  (WHO OSCI - World health Organization, Ordinal Scale for Clinical Improvement; 0=uninfected - 8=death)
Time Frame: 42 days
Population: All participants providing data at the relevant timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Participants
  Day 4 | 7 | 7
  Day 7: number analyzed (Participants) | 7 | 5
  Day 7 | 6 | 3
  Day 14: number analyzed (Participants) | 6 | 6
  Day 14 | 5 | 4
  Day 21: number analyzed (Participants) | 6 | 6
  Day 21 | 5 | 4
  Day 42: number analyzed (Participants) | 5 | 3
  Day 42 | 4 | 3

7. Secondary Outcome: Percentage of Participants Reporting Each Level of the WHO OSCI Score at Their Worst Post-baseline Day
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using percentage of participants reporting each level of the WHO OSCI score at their worst post-baseline day.
  (WHO OSCI - World health Organization, Ordinal Scale for Clinical Improvement; 0=uninfected - 8=death)
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Participants
  Score = 3 | 1 | 0
  Score = 4 | 4 | 7
  Score = 5 | 2 | 1
  Score = 6 | 0 | 1
  Score = 7 | 0 | 0
  Score = 8 | 0 | 0

8. Secondary Outcome: The Time in Days Spent at Each Participant's Worst Reported WHO OSCI Score (Excluding Death).
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using the time in days spent at each participant's worst reported WHO OSCI score (excluding death).
Time Frame: 42 days
Population: All participants providing data at the relevant timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Participants
  Score = 3; 1 day | 1 | 0
  Score = 3; 2-3 days | 0 | 0
  Score = 3; 4-7 days | 0 | 0
  Score = 3; >7 days | 0 | 0
  Score = 4; 1 day | 0 | 2
  Score = 4; 2-3 days | 2 | 3
  Score = 4; 4-7 days | 2 | 1
  Score = 4; >7 days | 0 | 1
  Score = 5: 1 day | 0 | 0
  Score = 5; 2-3 days | 1 | 0
  Score = 5; 4-7 days | 1 | 0
  Score = 5; >7days | 0 | 1
  Score = 6; 1 days | 0 | 0
  Score = 6; 2-3 days | 0 | 0
  Score = 6; 4-7 days | 0 | 0
  Score = 6; >7 days | 0 | 1
  Score = 7 | 0 | 0
  Score = 8 | 0 | 0

9. Secondary Outcome: Intubation and Mechanical-ventilation Free Survival
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using the intubation and mechanical-ventilation free survival, defined as the time in days from start of treatment to first occurrence of a WHO OSCI score of 6 or more.
  (WHO OSCI - World health Organization, Ordinal Scale for Clinical Improvement; 0=uninfected - 8=death)
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Participants
  Number of pts who died or required intubation/mechanical ventilation | 0 | 1
  Number of participants censored | 7 | 8

10. Secondary Outcome: Overall Survival
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using overall survival, defined as the time in days from start of treatment to death by any cause
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Participants
  Number of participants who died | 0 | 0
  Number of participants censored | 7 | 9

11. Secondary Outcome: Number of Days Requiring Oxygen Therapy
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using number of days requiring oxygen therapy
Time Frame: 42 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
days
  Days 1-14 | 6.9 (5.01) | 6.8 (4.52)
  Days 1-28 | 8.9 (9.30) | 8.8 (8.66)
  Days 1-42 | 10.9 (14.28) | 9 (9.22)

12. Secondary Outcome: Number of Days With Pyrexia
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using number of days with pyrexia ≥ 38C
Time Frame: 42 days
Population: All participants providing data within the relevant interval.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Days
  Days 1-14 | 0.1 (0.38) | 0.4 (0.73)
  Days 1-28 | 0.1 (0.38) | 0.4 (0.73)
  Days 1-42 | 0.1 (0.38) | 0.4 (0.73)

13. Secondary Outcome: Maximum Daily Temperature
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using maximum daily temperature
Time Frame: 42 days
Population: All participants providing data within the relevant interval.
Measure: Mean (Standard Deviation); unit: degress c
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
degress c
  Days 1-14 | 37.21 (0.414) | 37.32 (0.854)
  Days 1-28 | 37.21 (0.414) | 37.32 (0.854)
  Days 1-42 | 37.21 (0.414) | 37.32 (0.854)

14. Secondary Outcome: SpO2 Level
Description: The effect of 1815 on the development and severity of complications of COVID-19 infection will be measured using minimum and maximum SpO2 levels
Time Frame: 42 days
Population: All participants providing data within the relevant interval.
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
percentage of oxygen saturation
  Days 1-7 (min) | 92.3 (2.43) | 91.7 (2.18)
  Days 1-7 (max) | 96.0 (1.83) | 96.7 (2.50)
  Days 1-14 (min) | 92.0 (2.71) | 91.7 (2.18)
  Days 1-14 (max) | 96.0 (1.83) | 97.1 (2.37)
  Days 1-28 (min) | 92.0 (2.71) | 91.7 (2.18)
  Days 1-28 (max) | 96.0 (1.83) | 97.1 (2.37)
  Days 1-42 (min) | 92.0 (2.71) | 91.7 (2.18)
  Days 1-42 (max) | 96.6 (2.07) | 97.1 (2.37)

15. Secondary Outcome: Time to Discharge
Description: The effect of EDP1815 on length of hospitalization and recovery in participants with COVID-19 will be measured using time to discharge, defined as the time in days from start of treatment to first occurrence of a WHO OSCI score of 2 or less.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Participants
  Number of participants discharged | 6 | 6
  Number of participants who died | 0 | 0
  Number of participants censored | 1 | 3

16. Secondary Outcome: Time to Oxygen Saturation (SpO2) ≥94%
Description: The effect of EDP1815 on length of hospitalization and recovery in participants with COVID-19 will be measured using time to oxygen saturation (SpO2) ≥94% on room air without further requirement for oxygen therapy.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Participants
  Number of participants who achieved SpO2 >=94% without further requirement for oxygen therapy | 6 | 6
  Number of participants who died | 0 | 0
  Number of participants censored | 1 | 3

17. Secondary Outcome: Time to Recovery
Description: The effect of EDP1815 on length of hospitalization and recovery in participants with COVID-19 will be measured using time to recovery, defined as the time in days from symptom onset to alleviation of all COVID-19 symptoms.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Participants
  Number of participants who recovered | 4 | 4
  Number of participants who died | 0 | 0
  Number of participants censored | 3 | 5

18. Secondary Outcome: Number of Participants Experiencing AEs by Seriousness and Relationship to Treatment
Description: The safety and tolerability of EDP1815 in participants with COVID-19 will be measured using the number of participants experiencing AEs by relationship to treatment
Time Frame: 42 days
Population: The numbers analyzed only includes those participants who experienced adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Participants
  Acute Respiratory Distress Syndrome : Not related | 0 | 1
  Acute Respiratory Distress Syndrome : Related | 0 | 0
  Diarrhoea : Not related | 0 | 1
  Diarrhoea : Related | 0 | 0
  Abdominal distension : Not related | 0 | 1
  Abdominal distension : Related | 0 | 0
  Hypertension : Not related | 0 | 2
  Hypertension : Related | 0 | 0

19. Secondary Outcome: Incidence of Clinically Significant Abnormal Lab Parameters
Description: The safety and tolerability of EDP1815 in participants with COVID-19 will be measured using the number of participants experiencing clinically significant abnormal changes in safety lab parameters
Time Frame: 42 days
Population: Any clinically significant abnormal lab parameters were included as AEs.
Measure: Number; unit: number of participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
number of participants | 0 | 0

20. Secondary Outcome: Number of Participants Experiencing AEs by Seriousness and Relationship to Treatment
Description: The safety and tolerability of EDP1815 in participants with COVID-19 will be measured using the number of participants experiencing AEs by seriousness
Time Frame: 42 days
Population: Only serious AEs, AEs of CTCAE Grade 3 or above and AEs of special interest (all CTCAE grades) were documented and included in the summary.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | EDP1815
Number analyzed (Participants) | 7 | 9
Participants
  Acute Respiratory Distress Syndrome | 0 | 0
  Diarrhoea | 0 | 0
  Abdominal distension | 0 | 0
  Hypertension | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AE) and Serious Adverse Events (SAE) were documented from the point of informed consent up until 28 days post last administration of Investigational Medicinal Product (IMP), a maximum of up to 42 days post first administration of IMP.
Description: AEs were reported by the participant. Due to the nature of the patient population and disease, only SAEs and AEs of severe (CTCAE Grade 3) and potentially life threatening (CTCAE Grade 4) intensity were documented in the Case Report Form (CRF). AEs of mild (CTCAE Grade 1) or moderate (CTCAE Grade 2) intensity were documented in the medical notes. Adverse events relating to nausea, vomiting, diarrhoea, bloating and abdominal pain of any grade were recorded and assessed as an adverse events.
Arm/Group | Placebo | EDP1815
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/9
Other Adverse Events (participants affected / at risk) | 0/7 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | EDP1815 (N=9)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | EDP1815 (N=9)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT04488575/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT04488575/SAP_001.pdf